CLINICAL TRIAL: NCT07248072
Title: Effects of iPACK and Biceps Femoris Short Head (BiFeS) Blocks Combined With Adductor Canal Block on Quality of Recovery After Total Knee Arthroplasty: A Prospective, Randomized, Double-Blind Clinical Trial
Brief Title: Effect of iPACK and BiFeS Blocks on Quality of Recovery After Total Knee Arthroplasty
Acronym: BiFeS-TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Principal Investigator Ahmet Murat Yayık, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/769; 2025/2 (Other: Atatürk University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis; Postoperative Pain Management; Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Knee Replacement; Adductor Canal Block; iPACK Block; BiFeS Block; Regional Anesthesia; Postoperative Analgesia; QoR-15; Posterior Knee Pain; Ultrasound-Guided Nerve Block
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Single Person; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized, parallel-group design comparing iPACK and BiFeS blocks in combination with an adductor canal block.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will remain blinded to group allocation. The anesthesiologist performing the block procedures will not participate in postoperative assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor Canal Block + iPACK Block (Active Comparator): Participants in this arm will receive an ultrasound-guided adductor canal block (ACB) using 15 mL of 0.25% bupivacaine, followed by an iPACK (Interspace Between the Popliteal Artery and the Capsule of the posterior Knee) block with 25 mL of 0.25% bupivacaine. Blocks will be performed under sterile ultrasound guidance by an experienced anesthesiologist who will not participate in postoperative assessments. All patients will receive standardized spinal anesthesia and perioperative analgesia.
  Interventions: Procedure: Adductor Canal Block (ACB) Only; Procedure: IPACK block
- Adductor Canal Block + BiFeS Block (Experimental): Participants in this arm will receive an ultrasound-guided adductor canal block (ACB) using 15 mL of 0.25% bupivacaine, followed by a BiFeS (Biceps Femoris Short Head) block performed by injecting 25 mL of 0.25% bupivacaine into the potential space between the femur and the short head of the biceps femoris muscle. Procedures will be performed under sterile ultrasound guidance by an anesthesiologist not involved in postoperative assessments. All participants will receive standardized spinal anesthesia and perioperative analgesia.
  Interventions: Procedure: Adductor Canal Block (ACB) Only; Procedure: BiFeS Block

INTERVENTIONS:
Procedure: Adductor Canal Block (ACB) Only — An ultrasound-guided adductor canal block (ACB) will be performed using 15 mL of 0.25% bupivacaine. The probe will be placed on the proximal thigh to visualize the sartorius muscle and femoral artery. The needle will be advanced in-plane into the adductor canal, and correct placement will be confirmed with 2 mL saline before injection. This block aims to provide anterior knee analgesia while preserving quadriceps strength.
  Other Names: ACB
Procedure: IPACK block — The iPACK block will be performed by placing the ultrasound probe at the popliteal region to visualize the popliteal artery and posterior knee capsule. A needle will be advanced in-plane, and 25 mL of 0.25% bupivacaine will be injected between the artery and posterior capsule. This block targets posterior knee pain after total knee arthroplasty without causing motor block.
  Other Names: Interspace Between the Popliteal Artery and the Capsule Block; iPACK
  Arms: Adductor Canal Block + iPACK Block
Procedure: BiFeS Block — The BiFeS block will be performed with the ultrasound probe placed laterally to visualize the femur cortex and the long and short heads of the biceps femoris muscle. The needle will be advanced in-plane into the potential space between the femur and the short head of the biceps femoris. After confirming position with 2 mL saline, 25 mL of 0.25% bupivacaine will be injected. This block provides posterolateral knee analgesia with limited motor involvement.
  Other Names: Biceps Femoris Short Head Block; BiFeS
  Arms: Adductor Canal Block + BiFeS Block

SUMMARY:
This prospective, randomized, double-blind clinical trial aims to compare the effects of two different posterior knee analgesia techniques-iPACK block (Interspace Between the Popliteal Artery and the Capsule of the posterior Knee) and the Biceps Femoris Short Head (BiFeS) block-when combined with an adductor canal block (ACB) in patients undergoing elective unilateral total knee arthroplasty (TKA). Effective postoperative analgesia is essential for early mobilization, enhanced recovery, and patient satisfaction after TKA. Although ACB provides good anterior knee analgesia while preserving quadriceps strength, additional posterior knee analgesia is often required.

The iPACK block is a commonly used technique that targets the posterior knee capsule, whereas the newer BiFeS block aims to provide more selective posterolateral sensory blockade with potentially reduced risk of motor involvement. However, comparative clinical data between these two techniques are limited.

The primary objective of this study is to evaluate the difference between the iPACK and BiFeS blocks in terms of Quality of Recovery-15 (QoR-15) scores at 24 hours postoperatively. Secondary objectives include comparisons of postoperative pain scores, opioid consumption, time to first analgesic request, quadriceps and anterior tibialis muscle strength, functional test performance, time to mobilization, active range of motion, and the incidence of adverse events.

A total of 74 adult patients scheduled for elective unilateral TKA under spinal anesthesia will be randomized in a 1:1 ratio into two groups: ACB + iPACK block or ACB + BiFeS block. All blocks will be performed under ultrasound guidance by an experienced anesthesiologist. Outcome assessments will be conducted by blinded investigators. The study aims to provide high-quality clinical evidence regarding the effectiveness of the BiFeS block compared to the widely used iPACK technique.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind, parallel-group, single-center clinical trial designed to compare the effects of two posterior knee analgesia techniques-iPACK block and Biceps Femoris Short Head (BiFeS) block-when combined with an adductor canal block (ACB) on postoperative recovery outcomes following elective total knee arthroplasty (TKA). Postoperative pain after TKA is often severe and can limit early mobilization, delay rehabilitation, and negatively affect recovery. Multimodal analgesia strategies, including regional anesthesia techniques, play an essential role in optimizing postoperative outcomes.

The adductor canal block is widely used because it provides effective anterior knee analgesia while largely preserving quadriceps motor strength. However, it does not adequately address posterior knee pain. The iPACK block is frequently used to supplement ACB, providing analgesia to the posterior knee capsule by targeting the interspace between the popliteal artery and the posterior capsule. The BiFeS block is a newer regional anesthesia technique that involves injection between the femur and the short head of the biceps femoris muscle, targeting terminal sensory branches supplying the posterolateral knee. Cadaveric and early clinical data suggest that the BiFeS block may provide more selective posterior analgesia with limited spread to motor fibers, but comparative clinical data are scarce.

The primary objective of this study is to determine whether the combination of ACB + BiFeS block results in superior quality of recovery compared to ACB + iPACK block, as measured by the QoR-15 score at 24 hours postoperatively. Secondary outcomes include QoR-15 at 48 hours; pain scores at rest and during movement; total opioid consumption at 24 and 48 hours; time to first opioid request; quadriceps and anterior tibialis muscle strength; functional performance assessed using the Timed Up and Go (TUG) and Five Times Sit-to-Stand (FTSST) tests; active knee range of motion; time to first mobilization; and the incidence of adverse events such as nausea, vomiting, pruritus, sedation, neurological symptoms, local anesthetic systemic toxicity, and postoperative falls.

Eligible participants are adults aged 18-75 years undergoing elective primary unilateral TKA under spinal anesthesia, with an ASA physical status of I-III. Exclusion criteria include allergy to study medications, coagulopathy, anticoagulant therapy, severe cardiac, hepatic, or renal dysfunction, pre-existing neuropathic pain, infection at the injection site, neuromuscular disorders of the lower limb, pregnancy, or inability to cooperate with postoperative assessments. Written informed consent will be obtained from all participants. The study has received ethics approval from the Atatürk University Clinical Research Ethics Committee.

Participants will be randomized in a 1:1 ratio using computer-generated block randomization. Both patients and outcome assessors will remain blinded to group assignments. All block procedures will be performed under ultrasound guidance by an experienced anesthesiologist not involved in postoperative assessments. Standardized perioperative management will include spinal anesthesia with hyperbaric bupivacaine, perioperative non-opioid analgesics (paracetamol, dexketoprofen), antiemetic prophylaxis, and postoperative patient-controlled analgesia with fentanyl.

The sample size was calculated based on the minimal clinically important difference (MCID) for the QoR-15 score, assuming an effect size of 8 points, standard deviation of 10, power of 90%, and α = 0.05, resulting in 33 patients per group. Accounting for a 10% dropout rate, 74 patients will be enrolled.

Data will be analyzed using the intention-to-treat principle. Continuous variables will be compared with independent-samples t-tests or Mann-Whitney U tests based on distribution. Mixed-effects models will be used for repeated pain measurements. Categorical variables will be compared using chi-square or Fisher's exact tests. ANCOVA may be applied for adjusted analyses of QoR-15 outcomes.

This trial is expected to contribute important clinical evidence regarding the analgesic effectiveness, functional recovery benefits, and safety profile of the BiFeS block compared with the widely used iPACK block, helping guide postoperative analgesia strategies in total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Scheduled for elective primary unilateral total knee arthroplasty (TKA)
* Planned spinal anesthesia
* ASA physical status I-III
* Ability to understand study procedures and provide written informed consent

Exclusion Criteria:

* Known allergy or hypersensitivity to local anesthetics or other study medications
* Coagulopathy or current anticoagulant therapy
* Severe hepatic, renal, or cardiac failure
* History of neuropathic pain
* Infection at the site of proposed nerve block
* Pre-existing neuromuscular disorders in the lower extremities
* Inability to cooperate or refusal to participate in the study
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-15 (QoR-15) Score at 24 Hours | 24 hours postoperatively
  The Quality of Recovery-15 (QoR-15) questionnaire is a validated patient-reported outcome measure assessing overall postoperative recovery across domains such as pain, physical comfort, physical independence, psychological support, and emotional well-being. The total score ranges from 0 to 150, with higher scores indicating better recovery. The outcome compares 24-hour QoR-15 scores between the ACB + iPACK group and the ACB + BiFeS group.

SECONDARY OUTCOMES:
Quality of Recovery-15 (QoR-15) Score at 48 Hours | 48 hours postoperatively
  The QoR-15 questionnaire assesses multidimensional postoperative recovery, with scores ranging from 0 to 150 (higher scores indicate better recovery). This outcome compares 48-hour QoR-15 scores between the ACB + iPACK and ACB + BiFeS groups.
Pain Scores (VAS) at Rest and During Movement | 2, 4, 8, 12, 24, and 48 hours postoperatively
  Pain intensity will be evaluated using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain). Assessments will be performed at rest and during movement at predefined postoperative time points.
Opioid Consumption (Fentanyl PCA) | 24 and 48 hours postoperatively
  Total fentanyl consumption will be extracted from patient-controlled analgesia (PCA) device records, including total delivered dose and number of boluses.
Time to First Opioid Request | Up to 48 hours postoperatively
  The interval between the end of surgery and the patient's first demand for opioid analgesia via PCA will be recorded, indicating the duration of effective postoperative analgesia.
Quadriceps and Anterior Tibialis Muscle Strength | 4, 8, 12, 24, and 48 hours postoperatively
  Muscle strength will be assessed using standardized manual muscle testing (0-5 scale) for quadriceps and anterior tibialis muscles. Higher scores reflect greater strength.
Timed Up and Go (TUG) Test | Postoperative Day 1 and Day 2
  Functional mobility will be evaluated using the TUG test, which measures the time required for a participant to stand from a seated position, walk 3 meters, return, and sit down. Shorter times indicate better mobility.
Five Times Sit-to-Stand Test (FTSST) | Postoperative Day 1 and Day 2
  Lower extremity functional strength will be assessed by recording the time required to stand up and sit down five consecutive times. Faster performance reflects better function.
Active Range of Motion (Knee Flexion and Extension) | Postoperative Day 1 and Day 2
  Knee flexion and extension will be measured using a goniometer to assess active range of motion. Higher degrees indicate improved postoperative mobility.
Time to First Mobilization | Up to 48 hours postoperatively
  The time from arrival in the postoperative care unit to the patient's first successful mobilization (standing or walking with assistance) will be recorded.
Adverse Events and Complications | Up to 48 hours postoperatively
  Adverse events including nausea, vomiting, pruritus, sedation, falls, neurological symptoms, block-related complications, and signs of local anesthetic systemic toxicity (LAST) will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Murat Yayık, Principal Investigator, Principal Investigator — Ataturk University Department of Anesthesiology and Reanimation; Mehmet Akif YILMAZ, assistant doctor, Study Director — Ataturk University Department of Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive patient health information, and data confidentiality will be strictly maintained according to institutional ethical guidelines.

REFERENCES:
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Kilicaslan A, Tulgar S, Ahiskalioglu A, Aycan IO, Kekec AF, Arici AG, Kilic G, Sindel M. Ultrasound-guided biceps femoris short head block: a novel regional anesthesia technique for the posterolateral knee. Pain Med. 2025 Nov 1;26(11):726-732. doi: 10.1093/pm/pnaf068. PMID 40418224
- [Background] Sarikaya Ozel E, Taflan MG. Ultrasound-Guided Biceps Femoris Short Head Block for Posterolateral Knee Analgesia After Total Knee Arthroplasty: A Case Report. A A Pract. 2025 Sep 23;19(9):e02060. doi: 10.1213/XAA.0000000000002060. eCollection 2025 Sep 1. PMID 40985541
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Background] Grosu I, Lavand'homme P, Thienpont E. Pain after knee arthroplasty: an unresolved issue. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1744-58. doi: 10.1007/s00167-013-2750-2. Epub 2013 Nov 8. PMID 24201900
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Result] Myles PS, Myles DB, Galagher W, Chew C, MacDonald N, Dennis A. Minimal Clinically Important Difference for Three Quality of Recovery Scales. Anesthesiology. 2016 Jul;125(1):39-45. doi: 10.1097/ALN.0000000000001158. PMID 27159009
- [Result] Kertkiatkachorn W, Kampitak W, Tanavalee A, Ngarmukos S. Adductor Canal Block Combined With iPACK (Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee) Block vs Periarticular Injection for Analgesia After Total Knee Arthroplasty: A Randomized Noninferiority Trial. J Arthroplasty. 2021 Jan;36(1):122-129.e1. doi: 10.1016/j.arth.2020.06.086. Epub 2020 Jul 2. PMID 32694032
- [Result] Abdullah MA, Abu Elyazed MM, Mostafa SF. The Interspace Between Popliteal Artery and Posterior Capsule of the Knee (IPACK) Block in Knee Arthroplasty: A Prospective Randomized Trial. Pain Physician. 2022 May;25(3):E427-E433. PMID 35652772